CLINICAL TRIAL: NCT02684422
Title: TRI-STAR: Initial and Chronic MRSA Infection in CF (TRanslational Investigation of STaph. Aureus Resistance)
Brief Title: Initial and Chronic Methicillin Resistant Staphylococcus Aureus (MRSA) Infection in Cystic Fibrosis (CF)
Acronym: TRI-STAR
Status: Completed | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Other Study IDs: 15-0636
Record Dates: First submitted 2015-09-18; First posted 2016-02-18 (Estimated); Last update posted 2022-01-20 (Actual); Status verified 2022-01

CONDITIONS: Methicillin-Resistant Staphylococcus Aureus; Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — * Sputum
  * Blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cystic Fibrosis with MRSA infection: Cystic Fibrosis patients that are admitted to the hospital for IV therapy targeting MRSA will give a sputum sample and complete symptom diaries at the beginning and end of therapy. There will be no intervention administered.
  Inclusion criteria are ability to produce sputum and having a chronic i.e. > 2 years of positive respiratory cultures, MRSA CF lung infection.
  Interventions: Other: Intervention N/A. Observational study

INTERVENTIONS:
Other: Intervention N/A. Observational study — There are no interventions to the subjects other than collection of an expectorated sputum since this is an observational study; There are no study groups.See details per detailed study description.

SUMMARY:
This study aims to examine features of MRSA that are associated with chronic MRSA infection and bacterial persistence despite IV antibiotic therapy. Subjects are asked to expectorate sputum and complete CF symptom diaries both at beginning and end of IV therapy.

DETAILED DESCRIPTION:
This is an observational, translational study examined bacterial morphology and function pre- vs. post antibiotic therapy in patients with CF who experience a pulmonary exacerbation that requires IV antibiotics.

All clinical care is dictated by the treating physician(s).

Inclusion criteria:

1. Male or female with a confirmed diagnosis of CF (by sweat test and/or identification of 2 CF disease causing mutations).
2. Chronic infection with MRSA defined as having had MRSA positive respiratory cultures for > 1 year with > 50% of cultures being MRSA positive.
3. Being able to expectorate sputum on a consistent basis, i.e. also at the end of IV therapy 3A: starting April 2017 people with CF who cannot expectorate sputum can also participate if they will do two orapharyngeal swab cultures.
4. Having a pulmonary exacerbation defined for this protocol as the decision of the treating physician to start IV therapy in hospital or at home. Typically this occurs when there has been a >5% drop in FEV1 % predicted compared to the patient's baseline and increased respiratory symptoms.

   1. NOTE: Patients who had oral or inhaled antibiotics with or without MRSA activity but failed i.e. are changed to IV antibiotics are allowed to participate.

Exclusion criteria:

1. Presence / infection with B. cepacia genomovar III (B. cenocepacia)
2. Subjects who have undergone lung or liver transplant in the past (NOTE: patients listed for transplant are eligible)
3. Concomitant participation and/or use of an investigational drug within 30 days of this study. Concomitant observational studies are allowed with TRI-STAR

Sputum collection:

The subject will be asked to expectorate a sputum into a sterile specimen cup solely for this study. This may be a second sample after giving one for the clinical laboratory at start of therapy. The subject will be asked for a repeat sputum sample for the study at end of therapy.

Time point definition: A) Start of therapy sample: up to 3 days prior and up to 36 hours after the first dose of anti-MRSA antibiotic. B) End of therapy: no earlier than 36 hours prior to the last dose and up to one week after completion.

Collection of clinical information: Clinical information to be collected include: Demographics, age, CF genotype, anthropometrics; FEV1 FVC, FEF 25-75 in liter and % predicted per site specific reference values; all medications (routine and those started within 2 weeks and at time of admission/IV therapy).

CF daily Symptom score: Subject will be asked to complete the CF Symptom diary for the first and last 3 days of IV therapy. For subjects admitted to the hospital this will be administered by the RC for those at home the RC will call / e-mail them as reminder or do it with them per phone.

Spirometry at conclusion of therapy: Most patients have a follow-up clinic visit or are still in the hospital at time of completion of IV therapy and spirometry is part of routine clinical assessment. NOTE: Patients who would not have a clinic visit at end of therapy may be asked to return for spirometry and sputum sample solely for this study. If the subject agrees to this, reimbursement for travel will be allowed.

Laboratory Assays:

In vitro assays done on either banked isolates in Aim 1 or sputum samples / MRSA isolates from sputum include tests on bacterial fitness as growth under different conditions; antibiotic susceptibility assays; metabolic and virulence activity and genes, and mutator rates for sputum isolates. More details are provided in the grant application.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female with a confirmed diagnosis of CF (clinical features and positive sweat test and/or identification of 2 CF disease causing mutations).
2. At least 4 years of age or older.
3. Chronic infection with MRSA defined as having had MRSA positive respiratory cultures for > 1 year with ≥ 50% of cultures being MRSA positive e.g. 2/4 of the most recent cultures grew MRSA.
4. Being able to expectorate sputum on a consistent basis, i.e. also at the end of IV therapy.
5. Having a pulmonary exacerbation defined for this protocol as the decision of the treating physician to start IV therapy in hospital or at home. Typically this occurs when there has been a >5% drop in FEV1 % predicted compared to the patient's baseline and increased respiratory symptoms.

NOTE: Patients who had oral or inhaled antibiotics with or without MRSA activity but failed this outpatient therapy i.e. are changed to IV anti-MRSA antibiotics are allowed to participate.(Example: was on oral doxycycline and on admission changed to ceftaroline = eligible. On oral doxycycline that is continued on admission = not eligible).

* Patient enrollment should be prioritized to those receiving IV vancomycin or ceftaroline, with secondary consideration of patients who receive oral anti-MRSA therapy (TMP-SMX or a tetracycline derivative) that was initiated on hospital admission.
* Patients on linezolid will not be included as this medication is given orally and IV and may confound analyses.

Exclusion Criteria:

1. Presence / infection with B. cepacia genomovar III (=B. cenocepacia). Subjects who have undergone lung or liver transplant in the past (NOTE: patients listed for transplant are eligible)
2. Concomitant participation and/or use of an investigational drug within 30 days of this study.
3. Concomitant observational studies are allowed with TRI-STAR, if approved by the other study investigator or their proxy.

Ages: 4 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with a confirmed diagnosis of cystic fibrosis (CF), chronic MRSA who have a pulmonary exacerbation requiring IV therapy.
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2021-10 (Actual); Study Completion 2021-12 (Actual)

PRIMARY OUTCOMES:
Changes in presence of hypermutable MRSA isolates post-therapy compared to pre-therapy. | 2-3 weeks (course of IV antibiotics as determined by clinician)

SECONDARY OUTCOMES:
Other MRSA characteristics in sputum | 2 weeks (course of IV antibiotics)
  In vitro measures of MRSA fitness, antimicrobial susceptibilities, biofilm formation and exploratory in vitro bacterial assays.
Clinical improvement with therapy | 2-3 weeks (course of IV antibiotics)
  These measures for clinical improvement will be lung function and CF specific quality of life questionnaires.

CONTACTS AND LOCATIONS:
Overall Officials: Marianne S Muhlebach, MD, Principal Investigator — University of NC Chapel Hill, Dept Pediatrics
Locations (3):
- United States (3):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - University of Washington, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No
No plans to share individual patient data since the research study does not affect clinical outcomes, i.e. this is an observational study.